CLINICAL TRIAL: NCT06731114
Title: "Additional Effects of Sternocleidomastoid Release Along With Suboccipital Muscle Release in Management of Cervicogenic Headache'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/58
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups.one group will recieve conventional physical therapy including hot pack and tens for 10mins and suboccipital muscle release ( 3mins 3 reps) 9 mins .12 sessions in total where as group B will receive Sternocleidomastoid release for 5 mins along with suboccipital muscle release and conventional physical therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): On group A we will perform suboccipital muscle release (3 repititions 3 mins)9 minutes along with conventional physical therapy including TENS and hot pack for 10 mins 6 days a week for consective 2 weeks.
  Interventions: Procedure: Suboccipital muscle release; Procedure: Conventional physical therapy
- Group B (Experimental): On group B we will perform sternocleidomastoid release for 5 mins along with suboccipital muscle release and coventional physical therapy including TENS and hot pack for 10 mins 6 days a week for consective 2 weeks .
  Interventions: Procedure: Suboccipital muscle release; Procedure: Conventional physical therapy; Procedure: Sternocleidomastoid release

INTERVENTIONS:
Procedure: Suboccipital muscle release — Suboccipital muscle release.6 consecutive sessions for 2 weeks
  • Frequency:( 3mins 3 reps) 9 mins .12 sessions in total
Procedure: Conventional physical therapy — TENS and hot pack for 10 mins 6 days a week for consecutive 2 weeks
Procedure: Sternocleidomastoid release — Frequency: 5 mins of SCM release and 9 mins (3 mins 3 reps )of suboccipital release. 12 sessions in total.
  Arms: Group B

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the "Additional effects of sternocleidomastoid release along with suboccipital muscle release in management of cervicogenic headache".

DETAILED DESCRIPTION:
Cervicogenic headache is a common headache that causes disability and affects everyday activities. Headache related disorders are the second most common reason for years lived with disability all over the world. According to the latest International Headache Society model, cervicogenicheadache (CGH) is a secondary headache having C1-C2 dysfunction. There is marked limitation in cervical ROM specially rotation. Treatment indicated involves use of electrotherapy and thermal modalities. In addition, use of different manual therapy techniques are advocated to eliminate the root cause i.e. C1-C2 dysfunction treating. patients with cervicogenic headache are mostly presented with forward head posture and weak deep neck flexors which may excerbate the headache symptoms.Therefore The purpose of this study is to determine the ""Additional effects of sternocleidomastoid release along with suboccipital muscle release in management of cervicogenic headache

ELIGIBILITY:
Inclusion Criteria

* Participants will be included according to international classification of headache criteria which includes:
* Headache with neck stiffness
* Headache at least once a month in the last 3 months
* Headache with at least 4 score in Numeric Pain Rating Scale(NPRS)
* Unilateral headache with no shift of side
* Positive flexion rotation test (Rotation restriction is greater than 10 degrees)
* C1-C2 dysfunction
* Headache precipitated by sustained neck movements,myofacial trigger points palpation in neck
* Age group 18-45
* Both male and female

Exclusion Criteria:

* Cervical spondylosis
* Headache of non-cervical origin
* Dizziness or visual disturbance
* Cervical radiculopathy/ nerve root involvement/ disc herniation
* Cervical instability/ fracture
* Vertebrobasilar insufficiency
* Thoracic outlet syndrome
* Cervical spine surgery
* Cervical spondylolisthesis
* Spinal infection or tumors
* Osteoporosis
* meningitis
* subarachnoid hemorrhage

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks
  Pain will be measured on the basis of Numeric Pain Rating Scale score.
ROM | 2 weeks
  Cervical rotation will be measured through CROM device

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan